CLINICAL TRIAL: NCT02968043
Title: Application Research of Physiotherapeutic Scoliosis Specific Exercises in Adolescent Idiopathic Scoliosis
Brief Title: Efficacy of Physiotherapeutic Scoliosis Specific Exercises in Adolescent Idiopathic Scoliosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: Xinhua Hospital Chongming Branch (Unknown); Shanghai First Rehabilitation Hospital (Unknown); Shanghai Yangzhi Rehabilitation Hospital (Unknown); Shanghai Yangpu Daqiao Community Health Service Center (Unknown)
Responsible Party: Principal Investigator, Qing Du, Chief of Rehabilitation Department, Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: XH-16-041
Record Dates: First submitted 2016-11-11; First posted 2016-11-18 (Estimated); Last update posted 2020-11-03 (Actual); Status verified 2020-11

CONDITIONS: Scoliosis Idiopathic Adolescent
Keywords: physiotherapeutic scoliosis specific exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Active Comparator): Control group will perform generalised physiotherapy exercises for a 60-min period for 2 or 3 times a week under the guidance of experienced physiotherapists in an outpatient clinic and for a 20-min period per day under the supervision of the parents at home. Generalised physiotherapy exercises consist of stretching and strengthening activities.
  Interventions: Other: generalised physiotherapy exercises
- intervention group (Experimental): Intervention group will perform physiotherapeutic scoliosis specific exercises for a 60-min period for 2 or 3 times a week under the guidance of experienced physiotherapists with expertise in scoliosis in an outpatient clinic and for a 20-min period per day under the supervision of the parents at home. Physiotherapeutic scoliosis specific exercises consist of patient and family education, 3D self-correction, stabilizing exercises, balance training, breathing exercises, and training in activities of daily living.
  Interventions: Other: physiotherapeutic scoliosis specific exercises

INTERVENTIONS:
Other: physiotherapeutic scoliosis specific exercises — Physiotherapeutic scoliosis specific exercises (PSSE) is recommended as a first step in the treatment of AIS to halt curve progression by SOSORT guidelines. The PSSE program will be personalized according to the subject's curves characteristics. The program includes patient and family education, 3D self-correction, stabilizing exercises, balance training, breathing exercises, and training in activities of daily living. A physiatrist will give a detailed explanation of the aims, importance, methods, and procedure of an intervention to patients and their parents. Each subject will receive guidance from multiple physiotherapists to ensure that the treatment effects are the result of the protocol and not any particular physiotherapists.
  Arms: intervention group
Other: generalised physiotherapy exercises — Generalised physiotherapy exercises includes stretching and strengthening activities. Little evidence is in favor of generalised physiotherapy exercises. Each subject will receive guidance from multiple physiotherapists.
  Arms: control group

SUMMARY:
Adolescent idiopathic scoliosis (AIS) has a relatively high prevalence in adolescents. Exercise is the most common conservative therapy for mild AIS patients. There are increasing evidences suggesting that physiotherapeutic scoliosis specific exercise (PSSE) can halt the curve progression. Nevertheless, the evidence concerning PSSE is inadequate and low quality. The aim of this study is to identify the efficacy of PSSE on Cobb's angle, rotation angle, fall index, pulmonary function, bone quality, and health related quality-of-life (HRQoL) for mild AIS patients, and to promote PSSE's application in Shanghai.

Prior to inclusion, all subjects will be examined by the physiatrists. A parent of each subject will be asked to sign an informed consent form before the subject participate in the study.

Eligible subjects will be randomized by a 1:1 allocation ratio by computer either to the intervention group, in which they will perform PSSEs; or the control group, in which they will perform generalised physiotherapy exercises. All subjects will be assessed at the initial visit and 6 months. A multidimensional, comprehensive evaluation including aesthetic appearance, radiographic measurement, static balance test, pulmonary function test, bone quality, and HRQoL will be used.

DETAILED DESCRIPTION:
Adolescent idiopathic scoliosis (AIS) is a complex three-dimensional deformity of the spinal column, including scoliosis in the coronal plane, fixed rotation of the vertebral body and physiological curvature loss in the sagittal plane. AIS has a relatively high prevalence in adolescents. Exercise is the most common conservative therapy for mild AIS patients and has been widely used to reduce spinal deformity and halt curve progression. There are two kinds of exercises: generalised physiotherapy exercises and physiotherapeutic scoliosis specific exercise (PSSE). Little evidence is in favor of generalised physiotherapy exercises. There are increasing evidences suggesting that PSSE can halt the curve progression. Nevertheless, the evidence concerning PSSE is inadequate and low quality. Thus, the aim of this study is to identify the efficacy of PSSE on Cobb's angle, rotation angle, fall index, pulmonary function, bone quality, and health related quality-of-life (HRQoL) for mild AIS patients, and to promote PSSE's application in Shanghai.

The AIS patients will be recruited from and investigated at the Xinhua Hospital, Xinhua Hospital Chongming Branch, Shanghai First Rehabilitation Hospital, Shanghai Yangzhi Rehabilitation Hospital, and Shanghai Yangpu Daqiao Community Health Service Centre. Prior to inclusion, all subjects will be examined by the physiatrists. The subjects' height, weight, shoulder, chest, back and pelvic asymmetries, and the Adams forward bend test will be evaluated and recorded. The following information will be obtained for all subjects, including demographic data (for example, age and sex), menarche status for the girls, and family history. A parent of each subject will be asked to sign an informed consent form before the subject participate in the study.

Eligible subjects will be randomized by a 1:1 allocation ratio by computer either to the intervention group, in which they will perform PSSEs under the guidance of an experienced physiotherapist with expertise in scoliosis in an outpatient clinic; or the control group, in which they will perform generalised physiotherapy exercises. All subjects will receive the treatment as allocated and will be assessed at the initial visit and 6 months. A multidimensional, comprehensive evaluation including aesthetic appearance, radiographic measurement, static balance test, pulmonary function test, bone quality, and HRQoL will be used.

ELIGIBILITY:
Inclusion Criteria:

* patients who are consistent with the diagnosis of adolescent idiopathic scoliosis suggested by Scoliosis Research Society
* the largest Cobb angle of less than 20 degrees on whole spine posterior-anterior X-ray radiographs in a standing position
* 10 to 16 years old
* skeletal immaturity with Risser sign of <3

Exclusion Criteria:

* previous exercises or brace treatment history
* previous operation history of spine or lower extremities
* scoliosis caused by neuromuscular disorder, vertebral malformation, trauma, tumor, or other diseases
* having contraindications to exercises

Ages: 10 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 42 (Estimated)
Dates: Start 2017-02-13 (Actual); Primary Completion 2021-12-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Cobb's Angle at 6 months | up to 6 months
  Cobb's angle is the "gold standard" measurement on the frontal plane. The standing full spine posterior-anterior X-ray radiograph will be taken at the initial visit and 6 months later.

SECONDARY OUTCOMES:
Rotation Angle of Apical Vertebral | up to 6 months
  Rotation angle of apical vertebral will be measured by Nash Moe rotation at the initial visit and 6 months later.
Change from Baseline Fall Index at 6 months | up to 6 months
  Static balance test will be performed at the initial visit and 6 months later. Fall index will be caculated. Fall index scores from 0 to 100. The higher the fall index the higher the risk of fall.
Change from Baseline Forced Vital Capacity at 6 months | up to 6 months
  Pulmonary function test will be tested at the initial visit and 6 months later. Forced vital capacity will be measured.
Change from Baseline Forced Expiratory Volume in First Second at 6 months | up to 6 months
  Pulmonary function test will be tested at the initial visit and 6 months later. Forced expiratory volume in first second will be measured.
Change from Baseline Nondominant Radius Speed of Sound at 6 months | up to 6 months
  Bone quality will be measured using a quantitative ultrasound machine (Omnisense 7000P, Sunlight Medical Inc, Israel) at the initial visit and 6 months later. The quantitative ultrasound method can measure speed of sound (SOS) at the distal 1/3 of the radius by axial transmission. The measurement site is defined as the distal 1/3 of the radius. The mean of three measurements of the radius SOS is used for analysis.
Scores of Scoliosis Research Society-22 Questionnaire | up to 6 months
  Scoliosis Research Society-22 questionnaire (SRS-22) scores will be evaluated using the Chinese version of SRS-22 at the initial visit and 6 months later. All subjects will be required to complete SRS-22 independently. SRS-22 is a simple form of questionnaire to assess the HRQoL of AIS patients. It consists of 22 questions in 5 domains including functional activity, pain, self-image, psychological heath and satisfaction to treatment. Each question scores from 1 point (the lowest) to 5 (the highest). Each domain scores from 5 points to 25 points except for satisfaction to the treatment, which scores from 2 points to 10 points. Each domain is expressed as a mean value: the higher the score the better the outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Qing Du, Ph.D, Principal Investigator — Xin Hua Hospital Affiliated to Shanghai Jiao Tong University School of Medicine
Locations (2):
- China (2):
  - Xin Hua Hospital affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - Xinhua Hospital Chongming Branch, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No